# Statistical Analysis Plan

| Trial Short Title | MinimALL |
|---|---|
| Trial Full Title | iMagINg of chemotherapy-Induced Morphological and functional lung changes in childhood Acute Lymphoblastic Leukemia and Hodgkin's disease |
| Funding | Internal |
| Trial Principle Investigator | Dr. med. A. Karow<br>PD Dr. med. F. Knieling |
| Statistical Analysis Plan Authors | Dr. med. A. Karow PD Dr. med. F. Knieling Dr. med. A. Dierl |
| Document Version | 1.1 |
| Document Version Date | 11.12.2024 |
| NCT-Number | 06093334 |

# **Table of content**

| 1. | Version History | 2 |
|----|-----------------------|------|
| 2. | Project summary | 3 |
| 3. | Scientific background | 4 |
| 4. | Study aims | 5 |
| 5. | Target variables | 6 |
| 6. | Study design | 7 |
| 7. | Study population | 8 |
| 8. | Biometry | . 10 |
| 9. | Statistical Analysis | . 11 |

# 1. Version History

# Version

Version 1.1

## **Version date**

11.12.2024

# Protokollversionen

| Date | Version | Authors | Changes |
|------------|---------|-------------------|----------------------|
| 10.08.2023 | 1.0 | Dr. med. A. Karow | |
| | | PD Dr. med. F. | |
| | | Knieling | |
| | | Dr. med. A. Dierl | |
| 11.12.2024 | 1.1 | Dr. med. A. Karow | Addition of the NCT- |
| | | PD Dr. med. F. | Number |
| | | Knieling | |
| | | Dr. med. A. Dierl | |

## 2. Project summary

With increasing cure rates of childhood cancer there is growing recognition of late effects of treatments. However, there is a lack of non-invasive and child-friendly procedures that can indicate possible late damage. This study uses morphologic and free-breathing phase-resolved functional low-field (PREFUL) magnetic resonance imaging (MRI) to identify persistent pulmonary toxicity after treatment for childhood acute lymphoblastic leukemia (ALL), Hodgkin's disease (HD) and allogeneic stem cell transplantation.

#### 3. Scientific background

Currently, overall cure rates of therapy for childhood acute lymphoblastic leukemia (ALL) and Hodgkin's disease (HD) exceed 80% [1]. Apart from the development of supportive measures and novel targeted therapies, this success is still based largely on the optimized and riskadapted dosing and scheduling of conventional chemotherapeutic agents and addition of radiotherapy in patients with HD in case of suboptimal response. Even though, contemporary systemic and local treatment regimens are less intensive than previous therapies, they are still associated with diverse general and specific, acute and chronic organ toxicities such as cardiac dysfunction, osteonecrosis, neurocognitive impairment, and second malignant neoplasms [2]. With increasing cure rates has come growing recognition of such adverse late effects of treatment and a number of guidelines for long-term follow-up (LTFU) after childhood cancer therapy have been proposed [3]. During treatment and aftercare, however, only crude orienting investigations assessing organ function are foreseen by these recommendations and apart from physical examinations and laboratory analyses, echocardiography remains the only functional imaging measure routinely applied according to the current protocols for pediatric ALL and HD. It appears conceivable, that by such investigations, minor organ alterations could be missed and additional approaches comprising more sensitive structural or functional imaging would be essential to facilitate early recognition and possible timely management of developing still subclinical alterations.

We here hypothesize that morphologic and free-breathing phase-resolved functional low-field (PREFUL) MRI may identify persistent pulmonary toxicity after treatment for childhood ALL and HD, respectively. Therefore, we propose to perform a cross-sectional, prospective, single-center clinical pilot study using low-field MRI in children and adolescents during the first five years after the end of therapy. The results of this trial could contribute to the implementation of further investigation techniques in future standardized and structured LTFU care.

#### References

- 1. Erdmann F, Frederiksen LE, Bonaventure A, Mader L, Hasle H, Robison LL, et al. Childhood cancer: Survival, treatment modalities, late effects and improvements over time. Cancer Epidemiol. 2021;71(Pt B):101733. Epub 2020/05/29. doi: 10.1016/j.canep.2020.101733. PubMed PMID: 32461035.
- 2. Silverman LB. Balancing cure and long-term risks in acute lymphoblastic leukemia. Hematology Am Soc Hematol Educ Program. 2014;2014(1):190-7. Epub 2015/02/20. doi: 10.1182/asheducation-2014.1.190. PubMed PMID: 25696854.
- 3. Gebauer J, Baust K, Bardi E, Grabow D, Stein A, van der Pal HJ, et al. Guidelines for Long-Term Follow-Up after Childhood Cancer: Practical Implications for the Daily Work. Oncol Res Treat. 2020;43(3):61-9. Epub 2020/01/14. doi: 10.1159/000504200. PubMed PMID: 31931503.

### 4. Study aims

Determination of the frequency of morphologic and functional lung parenchymal changes using low-field magnetic resonance imaging

### **Hypotheses:**

- Lung parenchymal changes can be detected in pediatric and adolescent patients after completion of chemotherapy or chemotherapy and additional radiotherapy
- Patients with changes do not present with clinical symptoms

### **Primary Objective:**

- To determine the frequency of morphologic lung parenchymal changes using LF-MRI.

#### **Secondary Objectives:**

- To determine the frequency of functional lung parenchymal changes using LF-MRI.
- Determination of the anamnestic frequency of clinical respiratory symptoms

#### Study type

Prospective, monocentric, diagnostic study

# 5. Target variables

# **Primary target variables:**

| LF-MRT Changes of lung parenchyma |
|-----------------------------------|
|-----------------------------------|

# Secondary target variables:

| LF-MRT | Functional lung parameters (Ventilation |
|-------------------------|-------------------------------------------------|
| | match/mismatch, Perfusion |
| | match/mismatch, combined defects) |
| Cardiopulmonary testing | Oxygen uptake (VO <sub>2</sub> ) |
| | peak oxygen uptake (VO₂max) |
| | Respiratory exchange ratio (RER) |
| | Ventilatory anaerobic threshold (VT2) |
| | Carbon dioxide output (VCO <sub>2</sub> ) |
| | Heart rate (HR) |
| | Heart Rate Reserve (HRR) |
| | Breath rate at VAT |
| | Breath rate reserve (BRR) |
| | minute ventilation (VE) |
| | O <sub>2</sub> Pulse |
| | Heart rate variability (HRV) |
| | Exercise capacity (Borg Scale) |
| | Capillary blood gases and lactate |
| | At time 0 and after 6 months |
| Blood sample | Blood count*, Enterocytes*, Liver enzymes*, |
| | Retentionparamters* |
| Pulmonary tests | Lung function (VC%, FEV1%) |
| Clinical parameters | Age* |
| | Gender* |
| | Weight* |
| | Ethnicity* |
| | Time from therapy initiation/Interval until LF- |
| | MRI |
| | Current medication* |
| | Secondary diagnoses* |
| | Clinical examination* |

<sup>\*</sup>Standard procedures/parameters routinely available in follow-up care

# 6. Study design

# **Monocentric / multicentric**

This is a monocentric study

## Study arms: intervention/control

Patients (early and late effects) fulfilling the inclusion criteria will receive an MRI of the lungs and lung function testing

### Randomization

Randomization is not planned

# **Blinding**

Blinding to the study is not possible. Blinding of patients/subjects is not necessary

# 7. Study population

## In- and exclusion criteria

| Early therapeutic effects | Late therapeutic effects | Effects of hematopoietic |
|---|---|---|
| | | stem cell transplantation |
| Planned number of patients | | |
| N=10 ALL | N=10 ALL | N=10 |
| N=10 HD | N=10 HD | |
| | Inclusion criteria | |
| - Diagnosed acute | - Diagnosed acute | - Diagnosed acute |
| lymphatic leukemia | lymphatic leukemia | lymphatic leukemia |
| or Hodgkin's disease | or Hodgkin`s disease | - Completed |
| (HD) | (HD) | hematopoietic ste |
| - Completed induction | - Completed intensive | cell transplantation |
| therapy or | therapy or | - From 5 years to <18 |
| radiotherapy | radiotherapy | years |
| - From 5 years to <18 | - From 5 years to <18 | |
| years | years | |
| | Exclusion criteria | |
| - Pregnancy, Lactation | - Pregnancy, Lactation | - Pregnancy, Lactation |
| - Known pleural or | - Known pleural or | - Known pleural or |
| pericardial effusion | pericardial effusion | pericardial effusion |
| - Critical condition | - Critical condition | - Critical condition |
| (requiring respiratory | (requiring respiratory | (requiring respiratory |
| support, ventilation, | support, ventilation, | support, ventilation, |
| oxygen, shock, | oxygen, shock, | oxygen, shock, |
| symptomatic heart | symptomatic heart | symptomatic heart |
| failure) | failure) | failure) |
| - Marked thoracic | - Marked thoracic | - Marked thoracic |
| deformities/malforma | deformities/malforma | deformities/malforma |
| tions | tions | tions |
| - Previous lung | - Previous lung | - Previous lung |
| surgery | surgery | surgery |
| - Injuries that do not | - Injuries that do not | - Injuries that do not |
| allow physical stress | allow physical stress | allow physical stress |
| diagnostics | diagnostics | diagnostics |

| - Rejection of MRI | - Rejection of MRI | - Rejection of MRI |
|-----------------------|-----------------------|-----------------------|
| imaging | imaging | imaging |
| - General | - General | - General |
| contraindications for | contraindications for | contraindications for |
| MRI examinations | MRI examinations | MRI examinations |
| (e.g. electrical | (e.g. electrical | (e.g. electrical |
| implants such as | implants such as | implants such as |
| cardiac pacemakers | cardiac pacemakers | cardiac pacemakers |
| or perfusion pumps, | or perfusion pumps, | or perfusion pumps, |
| etc.) | etc.) | etc.) |

#### Recruitment channels and measures

Patients (and parents) will be informed about the possibility to participate in the study in public notices and announcements on the homepage of the hospital as well as when visiting the pediatric clinic for hematology and oncology (including its outpatient clinics). If patients and their parents are interested to participate, they will be fully informed about the aims and methods (especially about the scientific/explorative nature of the study), the benefits and risks, and the revocability of participation in the study before giving their consent prior to study initiation. Patients in childhood and adolescence are additionally informed and educated about the study and its procedure in an age-appropriate manner.

### 8. Biometry

Explorative, hypothesis-generating study

#### **Power calculation**

No power calculation was performed as part of a pilot study. So far, there are no reliable preliminary data/measurements or similar to have conclusions about the frequency of possible changes. Therefore, in the context of this pilot study, a N=10 per group (patients with ALL, patients with HD, and patients after allogeneic hematopoietic stem cell transplantation) is considered reasonable.

#### **Statistical Methodology**

Continuous variables will be reported as mean with standard deviation, categorical variables as numbers with percentages if necessary. The occurrence of MRI changes is reported as a percentage of the population. All analyses are performed using GraphPad Prism (version 7.00 or later, GraphPad Software, La Jolla, CA, USA), RStudio (version 1.1.456 or later, RStudio Inc., Boston, MA, USA), or IBM SPSS Statistics (version 24 or later, IBM Corp., Armonk, NY, USA).

### 9. Statistical Analysis

#### **Primary Objective:**

The occurrence of morphologic lung parenchymal changes is given as a percentage of the study sample.

#### **Secondary Objectives:**

To determine the anamnestic frequency of clinical respiratory symptoms, results are reported as a percentage of the study sample.

To test for differences in early versus late therapy-induced changes in functional MRI parameters (V/Q Mismatch) and results of Cardiopulmonary/pulmonary/myocardial testing, a nonparametric Mann-Whitney U test is used for pairwise comparisons. For the comparison of therapy-induced changes between different oncological diseases, a nonparametric Kruskal-Wallis test is performed. P < .05 is considered to indicate statistically significant difference in all analyses.